CLINICAL TRIAL: NCT00896038
Title: The Effect of NK1R Antagonism on Alcohol Craving and PTSD Symptoms in Alcohol Dependent Patients With PTSD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 090136; 09-AA-0136 (Other: NIHCC)
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Results first posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Alcoholism; Alcohol Dependence; Posttraumatic Stress Disorder
Keywords: Alcohol Dependence; Alcohol Treatment; Alcoholics; Alcoholism; Posttraumatic Stress Disorder; PTSD
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aprepitant (Experimental): Following a 1-week placebo lead-in period subjects were given 125 mg of Aprepitant orally daily for 21 days
  Interventions: Drug: Aprepitant
- Placebo (Placebo Comparator): Subjects received oral placebo during the 1-week placebo lead-in and then daily for 21 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aprepitant — Aprepitant is a neurokinin 1 receptor antagonist shown to have anti-stress actions in preclinical studies, and antidepressant efficacy in human clinical trials
  Other Names: Emend
  Arms: Aprepitant
Drug: Placebo — Non-active placebo
  Arms: Placebo

SUMMARY:
Objective:

Alcoholism is highly co-morbid with post traumatic stress disorder (PTSD). Since stress and negative affective states are major relapse triggering factors for alcohol use, the negative symptoms associated with PTSD are thought to promote alcohol dependence. Substance P, which is released in the amygdala in response to stress, acts at NK1 receptors (NK1Rs) to mediate behavioral stress responses. Blockade of the NK1R represents a novel approach for anti-stress actions. In a recent double blind, placebo controlled study involving detoxified anxious alcoholics, we found that NK1R antagonism decreased alcohol cravings, attenuated cortisol response to stress, and significantly decreased insula activation in response to negative sensory input. The present study is intended to expand the findings and determine whether the NK1R is a candidate target for treating alcohol dependent patients with PTSD.

Study Population:

On hundred twenty participants with PTSD and co-morbid alcohol dependence will be recruited and stratified by PTSD etiology (60 participants each with civilian and combat PTSD, resp). Within each stratum, the treatment groups will be balanced for sex using urn randomization. Stratification is indicated since civilian and combat-related PTSD can theoretically have a different pathophysiology. Civilians typically experience a single trauma exposure of invariably high magnitude, resulting in symptoms immediately. Combat-related PTSD typically results from multiple traumatic exposures over a prolonged period of time, of variable magnitude, and frequently with delayed emergence of symptoms.

Design:

Participants will be admitted to the National Institute on Alcohol Abuse and Alcoholism (NIAAA) research inpatient unit at the NIH Clinical Research Center (CRC) under protocol number 05-AA-0121 for assessment and treatment of people with alcohol drinking problems, which provides diagnostic assessments and standard withdrawal treatment if needed. Participants will enter into the present protocol once such treatment, if needed is completed. Following inclusion, all participants will receive 1 week of single blind placebo, and will then be randomized to double blind treatment with aprepitant or placebo. Randomized treatment will be for 3 weeks. Spontaneous cravings for alcohol, and ratings of psychopathology will be obtained twice weekly on the inpatient unit throughout the study. Cravings as well as endocrine and immune responses will also be assessed in a challenge session that combines a social stressor and exposure to physical alcohol cues. During the final week, three sessions utilizing scripts will be carried out, on separate days in counter-balanced order, exposing the participant to personalized trauma, alcohol-associated or neutral stimuli. Cravings as well as endocrine and immune responses will also be assessed during the script presentations. A functional magnetic resonance imaging (fMRI) session will be carried out last to assess responses to affective stimuli. Participants will remain hospitalized throughout the study, and will remain on the unit for a three day post-medication monitoring period.

Outcome Measures:

The primary outcome will be craving alcohol and changes in PTSD symptoms resulting from the script sessions. Secondary outcomes will include cravings and changes in PTSD symptoms resulting from the combined social stress-alcohol cure challenge session, spontaneous craving and PTSD symptoms during hospitalization, and brain responses on the fMRI session. Changes in PTSD symptoms and cravings for alcohol are intended to be surrogate markers for the overall effect of the drug treatment and are not intended to represent global improvement for either PTSD or alcoholism.

DETAILED DESCRIPTION:
Objective:

Alcoholism is highly co-morbid with post traumatic stress disorder (PTSD). Since stress and negative affective states are major relapse triggering factors for alcohol use, the negative symptoms associated with PTSD are thought to promote alcohol dependence. Substance P, which is released in the amygdala in response to stress, acts at NK1 receptors (NK1Rs) to mediate behavioral stress responses. Blockade of the NK1R represents a novel approach for anti-stress actions. In a recent double blind, placebo controlled study involving detoxified anxious alcoholics, we found that NK1R antagonism decreased alcohol cravings, attenuated cortisol response to stress, and significantly decreased insula activation in response to negative sensory input. The present study is intended to expand the findings and determine whether the NK1R is a candidate target for treating alcohol dependent patients with PTSD.

Study Population:

On hundred twenty participants with PTSD and co-morbid alcohol dependence will be recruited and stratified by PTSD etiology (60 participants each with civilian and combat PTSD, resp). Within each stratum, the treatment groups will be balanced for sex using urn randomization. Stratification is indicated since civilian and combat-related PTSD can theoretically have a different pathophysiology. Civilians typically experience a single trauma exposure of invariably high magnitude, resulting in symptoms immediately. Combat-related PTSD typically results from multiple traumatic exposures over a prolonged period of time, of variable magnitude, and frequently with delayed emergence of symptoms.

Design:

Participants will be admitted to the NlAAA research inpatient unit at the NIH Clinical Research Center (CRC) under protocol number 05-AA-0121 for assessment and treatment of people with alcohol drinking problems, which provides diagnostic assessments and standard withdrawal treatment if needed. Participants will enter into the present protocol once such treatment, if needed, is completed. Following inclusion, all participants will receive 1 week of single blind placebo, and will then be randomized to double blind treatment with aprepitant or placebo. Randomized treatment will be for approximately 3 weeks. Spontaneous cravings for alcohol, and ratings of psychopathology will be obtained twice weekly on the inpatient unit throughout the study. Cravings as well as endocrine and immune responses will also be assessed in a challenge session that combines a social stressor and exposure to physical alcohol cues. During the final week, three sessions utilizing scripts will be carried out, on separate days in counter-balanced order, exposing the participant to personalized trauma, alcohol associated or neutral stimuli. Cravings as well as endocrine and immune responses will also be assessed during the script presentations. An fMRI session will be carried out during week 4 to assess responses to affective stimuli. Participants will remain hospitalized throughout the study, and will remain on the unit for a three day post-medication monitoring period.

Outcome Measures:

The primary outcome will be change in craving for alcohol and changes in PTSD symptoms resulting from the script sessions. Secondary outcomes will include cravings and changes in PTSD symptoms resulting from the combined social stress-alcohol cue challenge session, spontaneous craving and PTSD symptoms during hospitalization, and brain responses on the fMRI session. Changes in PTSD symptoms and change in craving for alcohol are intended to be surrogate markers for the overall effect of the drug treatment and are not intended to represent global improvement for either PTSD or alcoholism.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Alcohol-dependent patients with a diagnosis of PTSD.
* Ages 21 - 50.
* Right-handed.
* Meet the Diagnostic and Statistical Manual (DSM)-IV diagnostic criteria for alcohol dependence (poly-substance abuse is common in younger alcohol-dependent patients and will not be exclusionary) and PTSD.
* Alcohol use within the last month.
* Females of childbearing potential must agree to use a reliable method of birth control during the study. Reliable methods of birth control include barrier methods such as diaphragms with contraceptive jelly, cervical caps with contraceptive jelly, condoms with contraceptive foam, or intrauterine devices; a partner with a vasectomy; or abstinence from intercourse. Hormonal contraceptives are not adequate in this study, because the study drug can render them less effective.

EXCLUSION CRITERIA:

* Individuals who present with complicated medical problems requiring intensive medical or diagnostic management.
* Individuals who are infected with the Human Immunodeficiency Virus (HIV).
* Individuals with serious neuro-psychiatric conditions which impair judgment or cognitive function to an extent that precludes them from providing informed consent or complying with treatment, such as psychotic illness or severe dementia (incompetent individuals).
* Individuals who are evaluated and judged by a board certified psychiatrist to be either severely depressed or an imminent risk for suicide, violence, or impulsive behavior, such as self-purging.
* Individuals who are unlikely or unable to complete the treatment program because they are likely to be incarcerated while on the protocol.
* Individuals who are required to receive treatment by a court of law or who are involuntarily committed to treatment.
* Pregnancy or lactation (negative pregnancy test required).
* A history of seizures, other than documented febrile seizures.
* Individuals currently using psychotropic medications will not be eligible for participation in the protocol if they are either unwilling or unable, for medical reasons, to be removed from their medication during hospitalization.
* Individuals in whom aprepitant is contraindicated because they take medications that can interact with this drug. Specifically, aprepitant should not be used concurrently with pimozide, terfenadine, astemizole, or cisapride. Dose-dependent inhibition of cytochrome P450 isoenzyme 3A4 (CYP3A4) by aprepitant could result in elevated plasma concentrations of these drugs, potentially causing serious or life-threatening reactions
* Inability or unwillingness to participate in an fMRI scan, including presence of metallic objects in the body that would interfere with the scan or pronounced claustrophobia.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2009-05; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David T George, M.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Andrews B, Brewin CR, Philpott R, Stewart L. Delayed-onset posttraumatic stress disorder: a systematic review of the evidence. Am J Psychiatry. 2007 Sep;164(9):1319-26. doi: 10.1176/appi.ajp.2007.06091491. PMID 17728415
- [Background] Asberg M, Schalling D. Construction of a new psychiatric rating instrument, the Comprehensive Psychopathological Rating Scale (CPRS). Prog Neuropsychopharmacol. 1979;3(4):405-12. doi: 10.1016/0364-7722(79)90055-9. PMID 400996
- [Background] Bergstrom M, Hargreaves RJ, Burns HD, Goldberg MR, Sciberras D, Reines SA, Petty KJ, Ogren M, Antoni G, Langstrom B, Eskola O, Scheinin M, Solin O, Majumdar AK, Constanzer ML, Battisti WP, Bradstreet TE, Gargano C, Hietala J. Human positron emission tomography studies of brain neurokinin 1 receptor occupancy by aprepitant. Biol Psychiatry. 2004 May 15;55(10):1007-12. doi: 10.1016/j.biopsych.2004.02.007. PMID 15121485
- [Derived] Kwako LE, Spagnolo PA, Schwandt ML, Thorsell A, George DT, Momenan R, Rio DE, Huestis M, Anizan S, Concheiro M, Sinha R, Heilig M. The corticotropin releasing hormone-1 (CRH1) receptor antagonist pexacerfont in alcohol dependence: a randomized controlled experimental medicine study. Neuropsychopharmacology. 2015 Mar 13;40(5):1053-63. doi: 10.1038/npp.2014.306. PMID 25409596

RESULTS

PARTICIPANT FLOW:
Groups:
- Aprepitant: Following a 1-week placebo lead-in period subjects were given 125 mg of Aprepitant daily for 21 days
- Placebo: Subjects received placebo during the 1-week placebo lead-in and then daily for 21 days
Period: Overall Study
Arm/Group | Aprepitant | Placebo
Started | 30 | 28
Completed | 26 | 27
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aprepitant | Placebo | Total
Number analyzed (Participants) | 30 | 28 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 28 | 58
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 16 | 15 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 30 | 26 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 14 | 28
  White | 16 | 12 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: Alcohol craving was measured using the Alcohol Urges Questionnaire (AUQ). The AUQ is an 8-item self-administered instrument that assesses craving for alcohol among alcohol users in the current context (i.e., right now). The score ranges from 8 (lowest craving value) to 56 (highest craving value).
Time Frame: 15 minutes prior to the beginning of stress script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 26 | 24
units on a scale | 11.9 (2.29) | 12.9 (2.39)

2. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 5 minutes after the beginning of stress script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 26 | 24
units on a scale | 20.9 (2.29) | 25.0 (2.38)

3. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 15 minutes after the beginning of stress script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 26 | 24
units on a scale | 19.2 (2.28) | 21.7 (2.39)

4. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 30 minutes after the beginning of stress script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 26 | 24
units on a scale | 18.0 (2.28) | 18.0 (2.39)

5. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 45 minutes after the beginning of stress script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 26 | 24
units on a scale | 18.1 (2.28) | 18.3 (2.38)

6. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 60 minutes after the beginning of stress script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 26 | 24
units on a scale | 15.9 (2.28) | 17.0 (2.38)

7. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 75 minutes after the beginning of stress script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 26 | 24
units on a scale | 15.9 (2.28) | 16.8 (2.38)

8. Primary Outcome: Alcohol Craving in Response to the Stress Script
Description: as for outcome 1
Time Frame: 90 minutes after the beginning of stress script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 26 | 24
units on a scale | 15.9 (2.28) | 14.1 (2.38)

9. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 15 minutes prior to the beginning of alcohol script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 26 | 24
units on a scale | 13.8 (2.05) | 14.0 (2.14)

10. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 5 minutes after the beginning of alcohol script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 26 | 24
units on a scale | 19.7 (2.05) | 20.7 (2.15)

11. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 15 minutes after the beginning of alcohol script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 26 | 24
units on a scale | 16.7 (2.05) | 16.3 (2.14)

12. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 30 minutes after the beginning of alcohol script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 26 | 24
units on a scale | 16.5 (2.05) | 14.4 (2.14)

13. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 45 minutes after the beginning of alcohol script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 26 | 24
units on a scale | 14.7 (2.05) | 15.1 (2.14)

14. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 60 minutes after the beginning of alcohol script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 26 | 24
units on a scale | 14.3 (2.05) | 14.4 (2.14)

15. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 75 minutes after the beginning of alcohol script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 26 | 24
units on a scale | 15.6 (2.05) | 13.6 (2.14)

16. Primary Outcome: Alcohol Craving in Response to the Alcohol Cue Script
Description: as for outcome 1
Time Frame: 90 minutes after the beginning of alcohol script presentation, which occurred on Day 25, 26, or 27 of the treatment period
Population: The analyses included only those subjects who completed all three script types (neutral, alcohol, stress)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 26 | 24
units on a scale | 14.8 (2.05) | 13.6 (2.14)

17. Primary Outcome: PTSD Total Symptom Severity Score
Description: PTSD total symptom severity was measured using the Clinician-Administered PTSD Scale (CAPS). This is a 30-item interview-based questionnaire that measures symptom severity during the past week. The total symptom severity score ranges from 0 (lowest symptom severity) to 136 (highest symptom severity).
Time Frame: Day 29 of the treatment period, 2 days after the final script presentation
Population: The analysis included subjects who completed the CAPS at both baseline (Day 1) and Day 29, and who had data for the baseline covariates used in the analysis
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Aprepitant | Placebo
Number analyzed (Participants) | 23 | 24
units on a scale | 53.0 (4.79) | 54.2 (4.66)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected biweekly throughout the 32 day inpatient stay
Arm/Group | Aprepitant | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/28
Other Adverse Events (participants affected / at risk) | 30/30 | 25/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aprepitant (N=30) | Placebo (N=28)
Constipation (Gastrointestinal disorders) | 14 | 8
Diarrhea (Gastrointestinal disorders) | 7 | 6
DryMouth (Gastrointestinal disorders) | 7 | 5
Flatulence (Gastrointestinal disorders) | 6 | 6
Nausea (Gastrointestinal disorders) | 9 | 11
Stomach or AbdominalAching (Gastrointestinal disorders) | 13 | 9
Fatigue or Weakness (General disorders) | 18 | 13
Irritability (General disorders) | 12 | 15
Nightmares (General disorders) | 2 | 1
Sleepiness (General disorders) | 2 | 0
Sweating (General disorders) | 8 | 5
Lack of Appetite (Metabolism and nutrition disorders) | 2 | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Dizziness (Nervous system disorders) | 7 | 6
Headaches (Nervous system disorders) | 18 | 18
Anxiety (Psychiatric disorders) | 0 | 4
Insomnia (Psychiatric disorders) | 2 | 2
Nervousness (Psychiatric disorders) | 10 | 9
Nightmares (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 2 | 1
SexualDysfunction (Reproductive system and breast disorders) | 3 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Itching (Skin and subcutaneous tissue disorders) | 2 | 2
Upset Stomach (Gastrointestinal disorders) | 9 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes